CLINICAL TRIAL: NCT06219655
Title: Extended Versus Limited Thoracoscopic Sympathectomy: Its Impact on Palmar and Plantar Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed emad, Lecturer of vascular surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.18.12.368.R1
Record Dates: First submitted 2024-01-04; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hyperhidrosis Due to Autonomic Dysregulation (Disorder)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended symathectomy (Active Comparator)
  Interventions: Procedure: thoracoscopic sympathectomy
- limited sympathectomy (Active Comparator)
  Interventions: Procedure: thoracoscopic sympathectomy

INTERVENTIONS:
Procedure: thoracoscopic sympathectomy — sympathectomy

SUMMARY:
Conclusions: In the context of palmar and plantar hyperhidrosis, extended thoracoscopic sympathectomy seemed to be preferred over limited thoracoscopic sympathectomy due to better overall outcomes and minimal time for hospital stays and Compensatory hyperhidrosis.

DETAILED DESCRIPTION:
ABSTRACT Objective: The aim was to carefully evaluate and compare the results of extended sympathectomy versus T3, T4, and T5 resection in cases of palmer, axillary, and planter hyperhidrosis as regards decreased sweating and recurrence rates.

Methods: This was a randomized controlled prospective trial conducted at the Department of Vascular Surgery Mansoura University Hospitals on a total of 120 patients with hyperhidrosis who were divided into two groups; group 1 who had undergone limited sympathectomy and group 2 who had undergone extended sympathectomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hyperhydrosis
* Able to take drugs
* Palmer and planter hyperhydrosis
* Age from 6-24 years
* Interfere with daily activities

Exclusion Criteria:

* Not fit for surgery
* Thyroid disease
* age less than 6 years
* Chest or cardiac problems

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
hyperhidrosis dryness of hands | from 2019-2023 over 4 years
  dryness of both hands and feet- difference in temperature hands and feet before and after-starch iodine test
dryness of both feet | from 2019-2023 over 4 years
  dryness of both hands and feet- difference in temperature hands and feet before and after-starch iodine test

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes